CLINICAL TRIAL: NCT00212082
Title: Gene Expression Profiles of Breast Cancer Treated With Sequential Adriamycin and Docetaxel in Relation to Tumor Responses
Brief Title: Gene Expression Profiles in Predicting Chemotherapy Response in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO B17/02
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; chemotherapy response; gene expression profiles; proteomics
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Docetaxel

INTERVENTIONS:
Drug: doxorubicin, docetaxel

SUMMARY:
We hypothesize that changes in tumor gene expression profiles vary in response to different sequences and types of chemotherapy, and that gene expression changes will correlate with tumor response. We are also looking to correlate drug pharmacokinetics and treatment toxicity with genotype of drug metabolizing enzymes and tranporters.Patients with metastatic breast cancer and who have measurable primary breast tumor will be randomized to one of two alternating sequences of adriamycin and docetaxel. Serial tumor biopsies and plasma samples will be obtained for gene expression and proteomic studies to identify biomarkers that will predict for chemotherapy response.

DETAILED DESCRIPTION:
Significant inter-individual variation exists in tumor response and chemotherapy toxicity because of unique tumor and patient factors. Individual drugs with distinct mechanisms of action may induce specific genomic and proteomic changes that may be used as predictor for response. We plan to study serial genomic and proteomic profiles in primary breast tumor treated with one of two sequences of alternating adriamycin (A) and docetaxel (T), A>T>A>T>A>T, or T>A>T>A>T>A, at 75mg/m2 3 weekly for each drug. Pharmacokinetic analysis of both drugs will be performed; amplified tumor RNA will be hybridized on Affymetrix® HG-U133+2 array; tumor proteins will be fractionated and profiled with ProteinChip® Array SELDI MS (Ciphergen). Tumor gene expression and proteomic changes will be correlated with treatment response to identify biomarkers that may predict chemotherapy sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Female, age > 18 years.
* Histologic or cytologic diagnosis of breast carcinoma.
* Stage II to IV breast cancer with measurable primary breast tumor, defined as palpable tumor with both diameters 2.0cm or greater as measured by caliper.
* Patients must not have received prior chemotherapy or hormonal therapy for the treatment of breast cancer.
* Karnofsky performance status of 70 or higher.
* Estimated life expectancy of at least 12 weeks.
* Adequate organ function including the following:

  - Bone marrow: White blood cells (WBC) >= 3.5 x 109/L Absolute neutrophil (segmented and bands) count (ANC) >= 1.5 x 109/L Platelets >= 100 x 109/L Haemoglobin >= 9g/dL

  - Hepatic: Bilirubin <= 1.5 x upper limit of normal (ULN), ALT or AST <= 2.5x ULN, (or <=5 X with liver metastases) Alkaline phosphatase <= 2.5x ULN.

  - Renal: creatinine <= 1.5x ULN
  * Cardiac:
  * Adequate cardiac function
* Signed informed consent from patient or legal representative.
* Patients with reproductive potential must use an approved contraceptive method if appropriate (eg, intrauterine device, birth control pills, or barrier device) during and for three months after the study. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

* Prior treatment for locally advanced or metastatic breast cancer.
* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia.
* Peripheral neuropathy of >= CTC grade 2.
* History of hypersensitivity to drugs formulated in Tween 80, the vehicle used for commercial docetaxel formulations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-04

PRIMARY OUTCOMES:
1. Evaluate the impact of adriamycin and docetaxel on tumor gene expression profiles.
2. Correlate overall tumor response with tumor gene expression profiles.

SECONDARY OUTCOMES:
To correlate adriamycin and docetaxel pharmacokinetics with:
1. Genetic polymorphisms of MDR-1, Cyp3A and GSTs.
2. Drug toxicity and tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Chin Lee, MD, Principal Investigator — Consultant
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Tan SH, Sapari NS, Miao H, Hartman M, Loh M, Chng WJ, Iau P, Buhari SA, Soong R, Lee SC. High-Throughput Mutation Profiling Changes before and 3 Weeks after Chemotherapy in Newly Diagnosed Breast Cancer Patients. PLoS One. 2015 Dec 2;10(12):e0142466. doi: 10.1371/journal.pone.0142466. eCollection 2015. PMID 26630576
- [Derived] Voon PJ, Yap HL, Ma CY, Lu F, Wong AL, Sapari NS, Soong R, Soh TI, Goh BC, Lee HS, Lee SC. Correlation of aldo-ketoreductase (AKR) 1C3 genetic variant with doxorubicin pharmacodynamics in Asian breast cancer patients. Br J Clin Pharmacol. 2013 Jun;75(6):1497-505. doi: 10.1111/bcp.12021. PMID 23116553
- [Derived] Chuah BY, Putti T, Salto-Tellez M, Charlton A, Iau P, Buhari SA, Wong CI, Tan SH, Wong AL, Chan CW, Goh BC, Lee SC. Serial changes in the expression of breast cancer-related proteins in response to neoadjuvant chemotherapy. Ann Oncol. 2011 Aug;22(8):1748-54. doi: 10.1093/annonc/mdq755. Epub 2011 Feb 25. PMID 21355070
- [Derived] Lim YW, Goh BC, Wang LZ, Tan SH, Chuah BYS, Lim SE, Iau P, Buhari SA, Chan CW, Sukri NB, Cordero MT, Soo R, Lee SC. Pharmacokinetics and pharmacodynamics of docetaxel with or without ketoconazole modulation in chemonaive breast cancer patients. Ann Oncol. 2010 Nov;21(11):2175-2182. doi: 10.1093/annonc/mdq230. Epub 2010 Apr 29. PMID 20430905
- [Derived] Lee SC, Xu X, Chng WJ, Watson M, Lim YW, Wong CI, Iau P, Sukri N, Lim SE, Yap HL, Buhari SA, Tan P, Guo J, Chuah B, McLeod HL, Goh BC. Post-treatment tumor gene expression signatures are more predictive of treatment outcomes than baseline signatures in breast cancer. Pharmacogenet Genomics. 2009 Nov;19(11):833-42. doi: 10.1097/FPC.0b013e328330a39f. PMID 19809382
- [Derived] Fan L, Goh BC, Wong CI, Sukri N, Lim SE, Tan SH, Guo JY, Lim R, Yap HL, Khoo YM, Iau P, Lee HS, Lee SC. Genotype of human carbonyl reductase CBR3 correlates with doxorubicin disposition and toxicity. Pharmacogenet Genomics. 2008 Jul;18(7):621-31. doi: 10.1097/FPC.0b013e328301a869. PMID 18551042